CLINICAL TRIAL: NCT02438176
Title: Comparison of Single Groin and Single Trans-septal Puncture and Conventional Bilateral Groin Puncture and Double Trans-septal Puncture in Catheter Ablation for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2015-0170
Record Dates: First submitted 2015-05-03; First posted 2015-05-08 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- single puncture group (Experimental): single trans-septal puncture
  Interventions: Procedure: single trans-septal puncture
- conventional group (Active Comparator): conventional bilateral groin puncture
  Interventions: Procedure: conventional bilateral groin puncture

INTERVENTIONS:
Procedure: single trans-septal puncture — The investigators will compare bilateral groin puncture AF ablation and single groin puncture AF ablation with 1:2 randomization.
  Arms: single puncture group
Procedure: conventional bilateral groin puncture — Bilateral groin puncture AF ablation is control procedure exactly same to routine AF ablation with double trans-septal puncture.
  Arms: conventional group

SUMMARY:
The purpose of this study is to compare single groin puncture and bilateral groin puncture during AF ablation procedure. The investigators will compare 1) the degree of patients' discomfort during hemostasis by questionaire, 2) procedure time, 3) complication rates, and 4) 1-year clinical recurrence rate of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients agreement of consent
2. Patients who age more than 19
3. patients who undergoing catheter ablation of atrial fibrillation
4. Patients who are not vascular disease

Exclusion Criteria:

1. patients who do not agree with study inclusion
2. persistent AF
3. Patients with vascular disease or venous anomaly
4. Patients with structural abnormality of the heart

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06-02; Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Patient's subjective discomfort | 6month after procedure

SECONDARY OUTCOMES:
Procedure time | 1day
Procedure related complication rate | 1 month after procedure
Long-term AF recurrence rate | 12 month after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea